CLINICAL TRIAL: NCT06136507
Title: An Open, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of Recombinant Human Coagulation Factor Ⅷ-Fc Fusion Protein (FRSW107) for Injection in Pediatric Patients With Severe Hemophilia A
Brief Title: Study of Efficacy and Safety of FRSW107 in Pediatric Patients With Severe Hemophilia A
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SS-107-III03
Record Dates: First submitted 2023-10-26; First posted 2023-11-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Severe Hemophilia A
Keywords: safetyeffectiveness; immunogenicity; effectiveness; Children; Teenagers
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The main test period and the extension period (Experimental): Group 1:≥6 years old and <12 years old; Group 2: <6 years old pediatric patients Preventive treatment: 25~50 is recommendedlU/kg, Q3D, can adjust the dose to 65 IU/kg based on the patient's response, and if necessary, the investigator can adjust the frequency of administration based on the clinical outcome of the subject (the occurrence of bleeding and its clinical manifestations) and the FVIII valley concentration.PK intensive blood collection will be performed for the PK subgroup at V1 (DO) and appropriate PK blood collection will be performed at other specified visit time points. After completion of ∠50EDs and 26 months of treatment, the original prophylactic regimen can be continued until 100EDs
  Interventions: Drug: FRSW107

INTERVENTIONS:
Drug: FRSW107 — experimental：Q3D.≥50EDs， Expansion phase：Q3D.100EDs
  Other Names: Recombinant Human Coagulation Factor Ⅷ，Fc Fusion Protein for Injection

SUMMARY:
This study was divided into four stages: screening period, main trial period, extension period and follow-up period.

In the main trial, both groups received FRSW107 prophylactic therapy. The recommended initial dose of prophylactic administration was 50 IU/kg, the dose range was 25 to 50 IU/kg, and the recommended frequency of administration was once every three days (Q3D). The dose range could be adjusted according to the patient's response. The main trial period was prophylaxis up to ≥50 exposure days (EDs) and ≥6 months.

The investigator may adjust the dose according to the clinical efficacy of the subjects (the occurrence of bleeding and its clinical manifestations) and the concentration of FⅧ valley according to the following principles.

If necessary, the investigator may adjust the dosing interval according to the clinical efficacy of the subject (the occurrence of bleeding and its clinical manifestations) and the concentration of FⅧ. Investigators are advised to inform sponsors or their research partners when adjusting doses and dosing intervals during prophylaxis.

After participants completed prophylaxis until ≥50EDs and ≥6 months, participants' willingness and investigator evaluation were used to decide whether to enter the extended trial. All subjects entering the extended phase continued with the original prophylactic regimen until 100EDs was dosed.

During the main trial period and the extended preventive treatment period, if the subjects have breakthrough bleeding events requiring treatment, hemostatic treatment of breakthrough bleeding with investigational drugs can be performed. The researchers can refer to the treatment guidance for different degrees of bleeding in Table 6-1. Taking into account the subject's prophylactic dose, severity of bleeding, site and extent of bleeding, clinical status, and previous PK results (if any), the investigator determines the appropriate dose to administer (recommended dose range: 25 to 50 IU/kg) and dosing times until the investigator assessed significant control of bleeding episodes (e.g. reduction of pain and swelling) or return to pre-bleeding activity. If the bleeding episode stops, the subject will continue with the same dose and frequency of prophylactic medication as before the bleeding episode.

ELIGIBILITY:
Inclusion Criteria:

1. Children <12 years old, male;
2. Weight >10kg;
3. clinically confirmed patients with severe hemophilia A (defined as confirmation at the time of screening or previous medical records: coagulation factor VI activity <1%);
4. Treated patients, that is, those who had previously received EVI treatment and met the following criteria: <6 years old patients who had been treated with coagulation factor VI for >50 exposure days (EDs250), and < 26 years old patients who had been treated with coagulation factor VI for >150 exposure days(> 150);
5. Normal prothrombin time (PT) or International normalized ratio (INR) <1.3;
6. At least 6 months of treatment and detailed records of bleeding events before screening;
7. The subject's legally authorized representative (i.e. guardian) fully understands and knows about this study and signs the informed consent. Children with the ability to give informed consent (≥8 years old) should be informed and sign the informed consent voluntarily;

Exclusion Criteria:

1. People who have been allergic to any component of EVI preparation (including but not limited to mouse or hamster protein or virus vaccine, gene recombination preparation containing mouse or hamster protein, etc.); Those who have had serious adverse reactions to previous vaccine injections or have not recovered from mild to moderate adverse reactions to vaccine injections; 2.Patients with hypersensitivity or anaphylaxis after injection of coagulation factor VI or Fc fusion protein products; 3. Positive factor VI inhibitor at screening (20.6 BU/mL), or previous history of factor VI inhibitor, or family history of inhibitor; 4.the screening results of von Willebrand factor (vWE) antigen were lower than the lower limit of normal value; 5. Severe anemia (hemoglobin <60g/L) at the time of screening; 6. Platelet count <100×10⁹ during screening /L; 7.abnormal liver function: alanine aminotransferase (ALT), or aspartate aminotransferase (AST) >3 times the upper limit of normal (ULN); Serum bilirubin (TBIL>3× ULN; 8. Patients with abnormal renal function: serum creatinine (SCr) >1.5×ULN or according toCreatinine clearance calculated by Cockcroft-Gault formula < 60 mL/min (CTCAE Level 1); 9. hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody, anti-human immunodeficiency virus antibody (Anti-HIV) and anti-treponema pallidum specific antibody (Anti-TP) test has one or more positive; 10. Patients with coagulation dysfunction other than hemophilia A; 11,.have other medical conditions that may increase the risk of bleeding or blood clots; 12. Have a known mental disorder that may affect trial compliance; 13. Patients who have used EV preparations of any standard half-life (e.g., Bekochi, Koyuki, Biinstop, Renjie, etc.) within 3 days or 5 half-lives prior to the first dose; Patients who have used any other half-life extension FVI preparations within 4 days or 5 half-lives prior to dosing (older at the time of retrieval); 14. Patients who have used emesezumab within 6 months prior to first dosing; 15. Severe cardiovascular and cerebrovascular disease, such as cerebral arteritis, moyamoya disease, stroke, viral myocarditis, endocarditis, endocardial fibroplasia, severe arrhythmia, congestive heart failure (New York Heart Association grade > III), uncontrolled hypertension, thromboembolic disease, and uncontrolled diabetes, occurred within 6 months prior to the first medication; 16. Patients who had used monoclonal antibody therapy, Fc fusion protein products, or intravenous immunoglobulin within 3 months before the first dose; 17.those who underwent major surgical procedures and transfusions of blood or blood components within 4 weeks prior to initial dosing, or who plan to undergo elective surgery (other than minor surgery such as tooth extraction) during the study treatment period; Those who underwent major surgical procedures and transfusions of blood or blood components within 4 weeks prior to initial dosing, or who plan to undergo elective surgery during the study treatment period; 18.patients with fever, active infection, allergies (such as allergic rhinitis, allergic asthma, allergic dermatitis, etc.) within 2 weeks prior to the first dose； 19.people with immune deficiency diseases or autoimmune diseases such as systemic lupus erythematosus, or have a history of organ transplantation or stem cell transplantation; Systemic immunomodulators (such as corticosteroids (>10mg/ day equivalent dose of prednisone), alpha-interferon, immunoglobulin, cyclophosphamide, cyclosporin, etc.) used within 14 days prior to the first administration or planned during the study period were allowed to use inhaled, nasal, ocular, intraarticular or topical corticosteroids; 20.patients who were treated with any anticoagulation (other than heparin sealing treatment) or platelet aggregation inhibitors within 7 days prior to initial administration or who required anticoagulation (other than heparin sealing treatment) or platelet aggregation inhibitors during study therapy; 21. Participants who have participated in other clinical trials within 1 month before screening; 22.had other serious medical conditions from which the researchers did not believe they could benefit; He suffered from severe skin disease, which interfered with the observation of local injection reaction.

23. Subjects deemed unsuitable by other investigators.

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2026-12-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ABR | 1year
  Number of bleeding during the treatment period/(Number of treatment days /365.25)

SECONDARY OUTCOMES:
AJBR | 1year
  annual rate of spontaneous joint bleeding and annual rate of traumatic joint bleeding
AE/ADR | 1year
  Frequency and severity of all AE/ADR and SAE/SAR
Incidence of positive FⅧ inhibitor | 1year
  Bethesda method improved by Nijmegen was adopted. Generally, the titers of 20.6 BU/ml were positive for two tests within 1-4 weeks. In addition to the screening period, FV1 inhibitor detection results 137/137Scheme number: SS-107-11103 ConfidentialVersion number: 4.0 Version Date: 07H August 2023The titer was 20.6 BU/ml, and retesting was scheduled within 1-4 weeks. At any visit, a minimum 72-hour FV1 washout period was required before collection of inhibitor test samples.
Cmax | 1year
  Cmax
Tmax | 1year
  Tmax
FⅧ activity | 1year
  FⅧ activity drops to 10%, 5%, 3%, 1% time

OTHER OUTCOMES:
Functional Independence Score in Hemophilia | 1 year
  FISH incorporates items that are perceived as important by persons with hemophilia, is performance based, and is relatively safe to perform.The higher the rating, the better
Pediatric Quality of Life Inventory | 1 year
  The higher the rating, the better

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Children's Hospital Affiliated to Chongqing Medical University, Chongqing
  - Guangzhou Women and Children Medical Center, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Affiliated Hospital of Guizhou Medical University, Guizhou
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou
  - Anhui Children's Hospital, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Nanjing Children's Hospital, Nanjing
  - Affiliated Hospital of Qingdao University, Qingdao
  - Shenzhen Children's Hospital, Shenzhen
  - Shanxi Children's Hospital, Taiyuan
  - Beijing Children's Hospital Affiliated to Capital Medical University, Tianjing
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No